CLINICAL TRIAL: NCT07353801
Title: The Efficacy and Safety of Oral Mini-pulse Dexamethasone in Active Non-segmental Vitiligo Within the Pediatric Age Group
Brief Title: Oral Mini Pulse Dexamethasone in Pediatric Vitiligo
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nanis Aleem Abdul Moneim Ragab, Associate professor Dermatology department Cairo University, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMPpedvitiligo
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Vitiligo
Keywords: oral mini pulse; vitiligo; pediatric; dexamethasone
MeSH Terms: conditions — Vitiligo | interventions — Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMP dexamethasone 2 consecutive days per week in a dose of 0.1mg/kg/day for 3 months (Experimental)
  Interventions: Drug: Dexamethasone (0.1 mg/kg)

INTERVENTIONS:
Drug: Dexamethasone (0.1 mg/kg) — patients will receive oral mini pulse dexamethasone 2 fixed consecutive days per week in a dose of 0.1mg/kg/day for a period of 3 months

SUMMARY:
The goal of this clinical trial is to learn if oral mini pulse (OMP) dexamethasone works to treat active vitiligo in children and also learn about the safety of this drug within this age group the main questions it aims to answer are does OMP halt activity in active vitiligo and what medical problems patients might experience while using the drug with special attention to linear growth. Researchers will give OMP dexamethasone to participating patients to see if the drug works to treat active vitiligo and whether it has any effect on linear growth. Participants will take OMP dexamethasone two fixed days per week for a period of 3 months. before starting treatment, patients will do baseline evaluation and investigations then monthly evaluation to monitor progress, report any side effects at the end of treatment period response to drug, lab values and growth will be evaluated then final evaluation of growth will be done after stoppage of drug.

DETAILED DESCRIPTION:
Background: Vitiligo is an autoimmune depigmenting skin disorder. Childhood Vitiligo (CV), defined as Vitiligo that begins before the age of 12 years, is common and may differ from post CV in terms of epidemiology, clinical picture, comorbidities and treatment options. Oral mini pulse (OMP) corticosteroids have been used successfully in both adults and children with active vitiligo. Pulsed regimens allow the achievement of the therapeutic outcome as well as better patient compliance while minimizing the adverse effects of daily steroids, However, its specific impact on linear growth in the pediatric population requires further evaluation. The aim of the current study is to evaluate the efficacy and safety of OMP dexamethasone in pediatric patients with active non-segmental vitiligo with special focus on linear growth.

Methodology: Male and female patients with active vitiligo defined as patients with Vitiligo disease activity score (VIDA) +3 and +4 patients with non-segmental vitiligo between 4-9 yrs will be included in the study. Baseline evaluation will include Vitiligo signs of activity score (VSAS) and Vitiligo area scoring index (VASI) scores, Routine lab investigations, HBA1c, cortisol am, ACTH am, blood pressure. Weight and height will be measured and plotted on WHO z score growth charts. Plain Xray of left hand and wrist for bone age will also be done. Patients will receive OMP dexamethasone in a dose of 0.1 mg/kg/day two consecutive days per week for 3 months. Topical treatment including topical betamethasone cream for body lesions and tacrolimus 0.1% cream for face lesions as well as puva sol /excimer laser will be allowed during the study. Patients will be monitored monthly to evaluate response and side effects. At the end of treatment period (3 months) the following parameters will be evaluated VSAS and VASI scores, weight and height plotted on WHO z scores growth charts. lab investigations including HBA1c, cortisol am and ACTH will be done one week after stoppage of treatment. 3 months after stoppage of treatment patients will be monitored for recurrence, weight and height will be measured and plotted on WHO z scores growth charts and bone age will be evaluated by plain Xray on left hand and wrist.

ELIGIBILITY:
Inclusion Criteria:

* Active (VIDA +3 & +4) non segmental vitiligo
* Age between 4-9yrs
* Males and Females
* Children with height measurements within the percentile range 5-95% of normal values for their age.

Exclusion Criteria:

* Segmental vitiligo.
* Stable vitiligo.
* History of endocrine disorders (growth hormone deficiency, thyroid disorders)
* Growth disorders (Turner's syndrome, Klinefelter's syndrome)
* Systemic diseases likely to affect growth (IBD, chronic renal failure)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The efficacy of dexamethasone in pediatric active non segmental vitiligo | 3 months
  Vitiligo signs of activity score (VSAS) will be evaluated and compared to baseline values. This scoring system ranges between (0-15). Zero means complete absence of clinical signs of activity. A decrease in the score at the end of the study compared to baseline values is considered an improvement (better outcome).
The effect of drug on bone age | 6 months
  Plain Xray left hand and wrist will be done 3 months after stoppage of drug and compared to baseline Xray.
The effect of drug on linear growth | 6 months
  The height of patients will be measured at baseline, at the end of treatment period and 3 months after stoppage of treatment. Height measurements will be done using a stadiometer and carefully read to the nearest 0.1 cm then height will be plotted on the WHO z-score growth charts.
The effect of drug on weight gain | 6 months
  Weight will be measured at baseline, at the end of treatment period and 3 months after stoppage of the drug. Weight will be measured using a digital scale and will be recorded to the nearest 0.1kg then measurements will be plotted on WHO z score growth charts.

SECONDARY OUTCOMES:
The effect of drug on HBA1C | 3 months
  HBA1c will be measured at the end of treatment period and compared to baseline values.
The incidence of adrenal suppression | 3 months
  Cortisol am and ACTH am will be measured at the end of treatment period and compared to baseline values
Incidence of patient reported corticosteroid side effects | 3 months
  patients will be followed up monthly during their treatment period, parents and patients will be questioned about the appearance of any of the following symptoms nausea, vomiting, epigastric pain, heart burn, increased appetite, weight gain and sleep disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Outpatient Clinic, Kasr al Ainy Teaching Hospital, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
I will share the deidentified data sheet of the results of the trial
Supporting Information: Study Protocol, SAP
Time Frame: 1 month after paper publication

REFERENCES:
- [Background] Nicolaidou E, Mastraftsi S, Tzanetakou V, Rigopoulos D. Childhood Vitiligo. Am J Clin Dermatol. 2019 Aug;20(4):515-526. doi: 10.1007/s40257-019-00430-0. PMID 30911977
- [Background] Lobato-Berezo A, March-Rodriguez A, Grimalt R, Rodriguez-Lomba E, Seto-Torrent N, Pujol RM, Ruiz-Villaverde R. Mini pulse corticosteroid therapy with oral dexamethasone for moderate to severe alopecia areata: A multicentric study. Dermatol Ther. 2022 Nov;35(11):e15806. doi: 10.1111/dth.15806. Epub 2022 Sep 16. PMID 36070222
- [Background] Sinha P, Sood A, Mukherjee B, Sinha A, Baveja S, Pathania V. Study to evaluate effect of oral mini pulse corticosteroid therapy for unstable vitiligo on hypothalamic pituitary adrenal axis suppression. Med J Armed Forces India. 2024 Dec;80(Suppl 1):S66-S72. doi: 10.1016/j.mjafi.2022.08.010. Epub 2022 Oct 22. PMID 39734899
- [Background] Majid I, Masood Q, Hassan I, Khan D, Chisti M. Childhood vitiligo: response to methylprednisolone oral minipulse therapy and topical fluticasone combination. Indian J Dermatol. 2009;54(2):124-7. doi: 10.4103/0019-5154.53185. PMID 20101306
- [Background] Radakovic-Fijan S, Furnsinn-Friedl AM, Honigsmann H, Tanew A. Oral dexamethasone pulse treatment for vitiligo. J Am Acad Dermatol. 2001 May;44(5):814-7. doi: 10.1067/mjd.2001.113475. PMID 11312430
- [Background] Kanwar AJ, Mahajan R, Parsad D. Low-dose oral mini-pulse dexamethasone therapy in progressive unstable vitiligo. J Cutan Med Surg. 2013 Jul-Aug;17(4):259-68. doi: 10.2310/7750.2013.12053. PMID 23815959
- [Background] Kanwar AJ, Dhar S, Dawn G. Oral minipulse therapy in vitiligo. Dermatology. 1995;190(3):251-2. doi: 10.1159/000246705. No abstract available. PMID 7599392
- [Background] Pasricha JS, Khaitan BK. Oral mini-pulse therapy with betamethasone in vitiligo patients having extensive or fast-spreading disease. Int J Dermatol. 1993 Oct;32(10):753-7. doi: 10.1111/j.1365-4362.1993.tb02754.x. PMID 8225724
- [Background] El Ghazaly, G. M., Albalat, W. M. and El Ghareeb, M. I. (2021) 'Use of oral mini pulse dexamethasone in vitiligo patients: Review article', Egyptian Journal of Hospital Medicine, 85(2), pp. 3909-3911. doi: 10.21608/ejhm.2021.205395.